CLINICAL TRIAL: NCT06224842
Title: A Phase Ib/II Clinical Study of Mitoxantrone Liposome and Azacitidine in the Treatment of Relapsed/Refractory Angioimmunoblastic T-cell Lymphoma
Brief Title: Clinical Study of Mitoxantrone Liposome and Azacitidine in the Treatment of R/R AITL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huijing Wu (Other)
Collaborators: Beijing Xisike Clinical Oncology Research Foundation (Unknown); CSPC Pharmaceutical Group (Unknown)
Responsible Party: Sponsor-Investigator, Huijing Wu, Deputy Chief Physician, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MitAITL
Record Dates: First submitted 2024-01-03; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Angioimmunoblastic T-cell Lymphoma
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mitoxantrone liposome and azacitidine treatment (Experimental): In the dose escalation phase, the mitoxantrone liposome will start at a dose of 16 mg/m^2 on day1 via intravenous infusion, combined with subcutaneous injection of azacitidine at a dose of 75 mg/m^2 on days 1-7, with each cycle lasting 4 weeks (28 days). Three predetermined dose groups for mitoxantrone liposome are 16, 18, and 20 mg/m^2. In the dose expansion phase, 10-20 cases will be included with the mitoxantrone liposome injection at the recommended phase II dose (RP2D) based on the results of the dose escalation phase.
  Interventions: Drug: mitoxantrone liposome 16 and azacitidine; Drug: mitoxantrone liposome 18 and azacitidine; Drug: mitoxantrone liposome 20 and azacitidine

INTERVENTIONS:
Drug: mitoxantrone liposome 16 and azacitidine — The mitoxantrone liposome will be intravenous infused at a dose of 16mg/m^2 on day1 , combined with subcutaneous injection of azacitidine at a dose of 75 mg/m^2 on days 1-7, with each cycle lasting 4 weeks (28 days).
Drug: mitoxantrone liposome 18 and azacitidine — The mitoxantrone liposome will be intravenous infused at a dose of 18mg/m^2 on day1 , combined with subcutaneous injection of azacitidine at a dose of 75 mg/m^2 on days 1-7, with each cycle lasting 4 weeks (28 days).
Drug: mitoxantrone liposome 20 and azacitidine — The mitoxantrone liposome will be intravenous infused at a dose of 20mg/m^2 on day1 , combined with subcutaneous injection of azacitidine at a dose of 75 mg/m^2 on days 1-7, with each cycle lasting 4 weeks (28 days).

SUMMARY:
This study is an open-label, single-arm Phase Ib/II clinical trial designed to evaluate the safety and efficacy of the combination therapy with mitoxantrone liposome and azacitidine in the treatment of relapsed/refractory angioimmunoblastic T-cell lymphoma(R/R AITL). The study includes two parts: a dose escalation phase and a dose expansion phase, each comprising screening, treatment, and follow-up periods. In the dose escalation phase, the mitoxantrone liposome injection will start at a dose of 16 mg/m^2 on day1, combined with subcutaneous injection of azacitidine at a dose of 75 mg/m^2 on days 1-7, with each cycle lasting 4 weeks (28 days). Three predetermined dose groups for mitoxantrone liposome are 16, 18, and 20 mg/m^2. In the dose expansion phase, 10-20 cases will be included with the mitoxantrone liposome injection at the recommended phase II dose (RP2D) based on the results of the dose escalation phase. After the treatment period, safety and survival information will be collected during the follow-up period. This study aims to comprehensively evaluate the safety and efficacy of mitoxantrone liposome in combination with azacitidine for the treatment of R/R AITL, exploring a combination therapy that offers higher survival benefits with limited adverse reactions and providing new therapeutic approaches for R/R AITL.

ELIGIBILITY:
Inclusion Criteria:

* The patient fully understands this study and voluntarily participates,willingly chooses to participate, and signs the informed consent form (ICF), expressing the willingness to comply with and having the capability to complete all trial procedures;
* Male or female patients aged 18 to 75(including 18 and 70 years old);
* ECOG score 0-2 points;
* Angioimmunoblastic T-cell lymphoma (AITL) confirmed by histopathology;
* Relapsed/refractory patients who have received at least first-line anthracyclines containing systematic therapy in the past. Relapsed lymphoma refers to lymphoma that relapses after obtaining a complete response (CR) or partial response(PR) after initial therapy.Refractory lymphoma is defined as progressive disease in the first chemotherapy cycle 2, or stable disease in the first chemotherapy cycle 4;
* There must be at least one measurable lesion that meets the Lugano2014 standard: a lymph node lesion, with a measurable lymph node length greater than 1.5cm in diameter; Non lymph node lesions, measurable extranodal lesions with a length diameter greater than 1.0cm;
* During patient screening, laboratory tests must meet the following requirements, and the patient should not have received any hematopoietic growth factors, platelet, or granulocyte transfusions within the 7 days prior to the hematological assessment during screening:

  1. neutrophil count ≥ 1.5 x 10^9/L, it can be relaxed to ≥ 1.0 x 10^9 /L in patients with bone marrow involvement;
  2. hemoglobin ≥ 90 g/L(without red blood cell transfusion within 14 days), it can be relaxed to ≥ 75 g/L in patients with bone marrow involvement;
  3. platelet count ≥ 75 x 10^9 /L, it can be relaxed to ≥ 50 x 10^9 /L in patients with bone marrow involvement;
  4. Total bilirubin ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver invasion);
  5. AST and ALT ≤ 2.5 times the upper limit of normal values ,≤ 5 times the upper limit of normal values for patients with liver invasion;
  6. Serum creatinine ≤ 1.5 times the upper limit of normal value; 8.Qualified patients of reproductive capability (both males and females) must agree to use a reliable contraceptive method with their partners during the trial and for at least 7 months after the last dose of medication. Female patients of childbearing age must have a negative blood pregnancy test within 7 days prior to enrollment.

Exclusion Criteria:

* Central nervous system (CNS) involvement or patients with hemophagocytic syndrome.
* History of allergy to similar drugs and excipients of the investigational drug.
* Patients with the following conditions in their history of prior antitumor therapy:

  1. Patients previously treated withMitoxantrone liposome in combination with Azacitidine (patients who have received either of the treatments, or those who have received both treatments sequentially, are eligible).
  2. Previous treatment with adriamycin or other anthracyclines, with a total cumulative dose of adriamycin ≥ 350 mg/m2 (conversion for other anthracycline-type drugs: 1 mg of daunorubicin/pirarubicin/epirubicin is equivalent to 0.5 mg of adriamycin, and 1 mg of idarubicin is equivalent to 2 mg of anthracycline).
  3. Receipt of cytotoxic chemotherapy, radiotherapy, targeted therapy within 4 weeks, immunomodulators (thalidomide, lenalidomide) within 3 weeks, or hormonal or herbal therapy for lymphoma within 2 weeks before the first dose of the investigational drug.
  4. Participation in other clinical trials and use of investigational drug treatment within 4 weeks before the first dose of the investigational drug.
  5. History of allogeneic hematopoietic stem cell transplantation or autologous hematopoietic stem cell transplantation within the past 6 months.
  6. Unresolved toxic reactions from prior anti-tumor therapy with toxicity persisting at > Grade 1, excluding alopecia and pigmentation.
  7. Impaired cardiac function or significant cardiac diseases, including but not limited to:

     1. Occurrence of myocardial infarction, congestive heart failure, or viral myocarditis within the past 6 months before screening;
     2. Symptomatic cardiac diseases requiring treatment intervention, such as unstable angina, arrhythmias, etc.;
     3. New York Heart Association (NYHA) functional class II-IV;
     4. Cardiac ejection fraction (EF) detected by echocardiography below 50% or below the lower limit of the laboratory reference range at the research center;
     5. Ongoing history of myocarditis;
     6. QTc > 450 milliseconds or congenital QT interval prolongation syndrome.
* Active hepatitis B (HBV surface antigen positive and HBV-DNA titer > 2000 IU/ml) or hepatitis C (HCV antibody positive and HCV-RNA titer higher than the upper limit of the normal range at the research center).
* History of severe autoimmune diseases, immunodeficiency diseases, including HIV antibody positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* History of malignant tumors within the past 5 years (excluding cured skin basal cell carcinoma and in situ cervical carcinoma).
* Underwent major surgery within the past 6 weeks or is expected to undergo major surgery during the study period.
* Uncontrolled hypertension (defined as blood pressure reaching stage 3 hypertension standards despite antihypertensive treatment, with systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 100 mmHg), or type 2 diabetes patients whose blood pressure cannot be controlled with oral hypoglycemic drugs and insulin therapy.
* Active bleeding history within the past 3 months before screening.
* History of mental illness or abuse and dependence on psychiatric drugs.
* Pregnant or lactating women.
* Other situations deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 2 year.
  The incidence and severity of treatment-emergent adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 2 year.
  the percentage of patients who achieve complete response or partial response.
Progression-Free Survival(PFS) | Through study completion, an average of 2 year.
  The time from the initiation of treatment until disease progression.
Overall Survival(OS) | Through study completion, an average of 2 year.
  The time from the start of treatment until the patient's death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Wu, Principal Investigator — Hubei Cancer Hospital
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No